CLINICAL TRIAL: NCT00960310
Title: Randomized, Open-Label, 1-Way Parallel, Bioequivalence Study of Bicalutamide 50 mg Tablet and Casodex (Reference) Following a 50 mg Dose in Healthy Subjects Under Fed Conditions.
Brief Title: Relative Bioavailability Study of Bicalutamide 50 mg Tablet and Casodex Following a 50 mg Dose in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60111
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-08

CONDITIONS: Prostate Cancer; Hirsutism
Keywords: Treatment
MeSH Terms: conditions — Prostatic Neoplasms; Hirsutism | interventions — bicalutamide

ARMS (2):
- 1 (Experimental): Bicalutamide 50 mg Film-Coated Tablets (Sandoz Inc., USA)
  Interventions: Drug: Bicalutamide 50 mg Film-Coated Tablets (Sandoz Inc., USA)
- 2 (Active Comparator): Bicalutamide 50 mg Film-Coated Tablets (Casodex) (Astrazeneca Pharmaceutical LP, USA)
  Interventions: Drug: Bicalutamide 50 mg Film-Coated Tablets (Casodex) (Astrazeneca Pharmaceutical LP, USA)

INTERVENTIONS:
Drug: Bicalutamide 50 mg Film-Coated Tablets (Sandoz Inc., USA)
  Arms: 1
Drug: Bicalutamide 50 mg Film-Coated Tablets (Casodex) (Astrazeneca Pharmaceutical LP, USA)
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the relative bioavailability of Bicalutamide 50 mg tablet and Casodex following a 50 mg dose in healthy subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — Anapharm